CLINICAL TRIAL: NCT06870877
Title: Neuropathic Pain and Traditional Medicine Syndromes in Herpes Zoster: a Cross-Sectional Study Conducted At Le Van Thinh Hospital, Vietnam
Brief Title: Neuropathic Pain and Traditional Medicine Syndromes in Herpes Zoster: a Cross-Sectional Study
Status: Not yet recruiting | Type: Observational
Sponsor: Do Thanh Sang (Other)
Responsible Party: Sponsor-Investigator, Do Thanh Sang, University of Medicine and Pharmacy at Ho Chi Minh City, University of Medicine and Pharmacy at Ho Chi Minh City
Organization: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Other Study IDs: 78/HĐĐĐ-ĐHYD
Record Dates: First submitted 2025-02-28; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-01

CONDITIONS: Herpes Zoster (HZ); Traditional Chinese Medicine (TCM)
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study investigates the relationship between neuropathic pain characteristics and Traditional Chinese Medicine (TCM) syndromes in patients with Herpes Zoster (HZ). The study aims to integrate objective pain assessment tools, such as the Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) scale, with TCM diagnostic classifications to enhance individualized treatment strategies. Conducted at Le Van Thinh Hospital, Vietnam, this cross-sectional study includes 80 HZ patients, assessing their pain levels and corresponding TCM syndromes. The findings will contribute to a more comprehensive approach to pain management in Herpes Zoster.

DETAILED DESCRIPTION:
This study is a cross-sectional and case series study conducted at Le Van Thinh Hospital, Ho Chi Minh City, Vietnam, between January and June 2024. It aims to evaluate the correlation between neuropathic pain characteristics and Traditional Chinese Medicine (TCM) syndromes in patients with Herpes Zoster (HZ). The study includes 80 participants diagnosed with HZ, whose pain severity is assessed using the Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) scale. The participants are classified into TCM syndromes based on standard diagnostic criteria, including Liver Meridian Depression and Heat Syndrome (LMD), Spleen Deficiency and Dampness Retention Syndrome (SDA), and Qi Stagnation and Blood Stasis Syndrome (QSA).

The primary objectives of the study are:

To determine the prevalence of different TCM syndromes in HZ patients. To analyze the correlation between LANSS scores and specific TCM syndromes. To provide insights into the integration of objective neuropathic pain assessment tools with traditional diagnostic frameworks.

Data collection includes demographic characteristics, medical history, pain characteristics, TCM diagnostic features, and clinical examination results. Statistical analyses include correlation tests and multinomial logistic regression to assess the relationship between LANSS pain scores and TCM syndromes.

The study findings will contribute to a better understanding of the relationship between neuropathic pain and TCM syndromes in Herpes Zoster. The results may help refine diagnostic approaches and optimize integrative treatment strategies for pain management in patients with HZ.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years
* Clinically diagnosed with Herpes Zoster (HZ) based on European Consensus Guidelines
* Experiencing neuropathic pain associated with HZ
* Willing to provide informed consent

Exclusion Criteria:

* History of chronic pain conditions unrelated to HZ
* Receiving immunosuppressive therapy or diagnosed with immunodeficiency disorders
* Patients who had already received antiviral or analgesic treatment before evaluation
* Patients unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of 80 adult patients diagnosed with Herpes Zoster (shingles) who presented at Le Van Thinh Hospital, Ho Chi Minh City, Vietnam. These patients were experiencing neuropathic pain and were assessed using the Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) scale. Participants were classified into Traditional Chinese Medicine (TCM) syndromes based on diagnostic criteria
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2025-05-12 (Estimated); Study Completion 2025-05-12 (Estimated)

PRIMARY OUTCOMES:
Neuropathic Pain Severity in Herpes Zoster Patients | Baseline (Day 1)
  Measured using the Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) pain scale. LANSS scores will be used to determine the severity of neuropathic pain in study participants.

SECONDARY OUTCOMES:
Correlation Between Neuropathic Pain and Traditional Medicine Syndromes | Baseline (Day 1).
  Analysis of LANSS scores and their association with Traditional Chinese Medicine (TCM) syndromes (Liver Meridian Depression and Heat Syndrome, Spleen Deficiency and Dampness Retention Syndrome, and Qi Stagnation and Blood Stasis Syndrome) using multinomial logistic regression.

CONTACTS AND LOCATIONS:
Locations (1):
- Le Van Thinh Hospital, Ho Chi Minh City, Viet Nam, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided